CLINICAL TRIAL: NCT06874140
Title: Biomarkers and Potential Mechanisms of Chinese Medicine Compound (Chuanhong Zhongfeng Capsule) in the Treatment of Acute Cerebral Infarction
Brief Title: Proteomic Study of Chuanhong Zhongfeng Capsule in the Treatment of ACI
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yingyue Ding (Other)
Responsible Party: Sponsor-Investigator, Yingyue Ding, Attending physician of the Department of Encephalopathy, Affiliated Hospital of Changchun University of Chinese Medicine
Organization: Affiliated Hospital of Changchun University of Chinese Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CCZYFYKYLL2023; 2022JC046 (Other Grant/Funding Number: Jilin Provincial Health Commission)
Record Dates: First submitted 2025-02-26; First posted 2025-03-13 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Chuanhong Zhongfeng capsule (Experimental): Basic treatment (refer to China Acute Ischemic Stroke Diagnosis and Treatment Guidelines 2018) + Chuanhong Zhongfeng capsule
  Interventions: Drug: Chuanhong Zhongfeng capsule
- control (Active Comparator): Basic treatment (refer to Chinese Guidelines for the Diagnosis and Treatment of Acute Ischemic Stroke 2018)
  Interventions: Drug: Chuanhong Zhongfeng capsule

INTERVENTIONS:
Drug: Chuanhong Zhongfeng capsule — Basic treatment (refer to China Acute Ischemic Stroke Diagnosis and Treatment Guidelines 2018) + Chuanhong Zhongfeng capsule

SUMMARY:
Acute cerebral infarction is characterized by high disability rate and high recurrence rate, which poses a great threat to the life and health of the nation. Proteomics technology is a holistic and comprehensive understanding of disease mechanism, cell metabolism and other processes at the protein level. The correlation between acute cerebral infarction and proteomics has become a hot spot of clinical and basic research in recent years. Chuanhong Zhongfeng capsule was developed by Ren Jixue, a master of national medicine, and clinical studies have confirmed that it not only promotes the recovery of neurological function in patients with cerebral infarction, reduces the disability rate, but also improves the long-term prognosis, but its mechanism of action and its target are still unclear. In the present study, we applied 4D Label-free proteomics technology and PRM technology to study for the first time the mechanism of action and potential targets of Chuanhong Zhongfeng Capsule in the treatment of acute cerebral infarction, which will provide a direction for the study of traditional Chinese medicine compounding for the prevention and treatment of cerebral infarction.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the diagnostic criteria for ischemic stroke in the Chinese Guidelines for Diagnosis and Treatment of Ischemic Stroke in the Acute Phase 2018.
2. Meet the diagnostic criteria for ischemic stroke in Chinese medicine.
3. Within 2 weeks of acute onset of ischemic stroke.
4. 4 ≤ NIHSS score <15.
5. Age 40-80 years old. -

Exclusion Criteria:

1. Diagnosis of hemorrhage or other pathological brain disorders based on head CT or MRI;
2. Allergic individuals, those who are allergic to the test medication or the associated medicinal flavors or components thereof;
3. Age <40 years or >80 years;
4. Those with severe liver or kidney function impairment. -

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Explore protein expression levels, post-translational modifications, protein-protein interactions, and obtain protein-level insights into disease mechanisms and disease biomarkers. | 14 day
  The study focused on identifying unique differential proteins in ACI patients treated with CHZF Capsule. Mass spectrometry analysis was performed using 4D label-free proteome quantification technology to identify differential proteins between the groups. Functional enrichment analysis, including GO classification and KEGG pathway analysis, was conducted to determine enrichment trends related to differential proteins. Hierarchical clustering was employed to identify relevant pathways enriched in each group based on P-values from the enrichment analysis. The STRING (v.11.5) protein interactions network database was utilized to obtain differential protein interactions, corresponding target proteins, and major related pathways. PRM was subsequently applied to validate the selected target proteins. Finally, chord diagrams and ROC curves were plotted for visualization and analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Changchun, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: ICF

REFERENCES:
- [Derived] Ding Y, Yao J, Wang X, Liu L, Niu P, Ma H, Zhang L, Wang X, Yang H, Zhao D, Nan H, Wang Y. Biomarkers and potential mechanisms of Chinese medicine compound (Chuanhong Zhongfeng Capsule) in the treatment of acute cerebral infarction. Phytomedicine. 2025 Sep;145:156955. doi: 10.1016/j.phymed.2025.156955. Epub 2025 Jun 11. PMID 40517620

DOCUMENTS (2):
  • Statistical Analysis Plan (2023-04-27): https://cdn.clinicaltrials.gov/large-docs/40/NCT06874140/SAP_000.pdf
  • Informed Consent Form (2023-04-27): https://cdn.clinicaltrials.gov/large-docs/40/NCT06874140/ICF_001.pdf